CLINICAL TRIAL: NCT06471062
Title: Transit Time Flow Measurement in Coronary Surgery: The Mutual Influence of Collateral Flow Between Different Coronary Territories on Parameter Metrics
Brief Title: Transit Time Flow Measurement in Coronary Surgery
Acronym: COLLATERAL
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Federico Cammertoni, Doctor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 6646
Record Dates: First submitted 2024-05-28; First posted 2024-06-24 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Coronary Artery Disease; Coronary Stenosis; Coronary Bypass Graft Stenosis
Keywords: coronary artery bypass; Transit Time Flowmetry; Intraoperative epicardial high-frequency ultrasound (HFUS); Coronary anastomosis patency
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Transit-time flowmetry (TTFM) allows grafts quality control during coronary artery bypass surgery by measuring the flow volume through them.

To date, many studies have deeply studied the predictive role on the graft outcomes of the various flowmetry-derived parameters. One of the least investigated aspects, however, is the mutual influence that two newly realized grafts can have. This possibility would be related to the presence of a more or less developed collateral circulation between the bypassed territories.

The purpose of this study is to assess whether a graft for a territory different than that provided by the left anterior descending artery (LAD) may affect the functionality (measured through flowmetry) of the left internal mammary artery - LAD graft.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years;
* informed consent acquired and registered;
* patients who undergo coronary artery bypass grafting (with or without cardiopulmonary bypass);
* patients with stable angina, unstable angina or acute coronary syndrome without elevation of the ST tract (NSTEMI)

Exclusion Criteria:

* patients unable to give informed consent;
* patients undergoing emergency surgery;
* patients in unstable haemodynamic conditions or in need of pharmacological or mechanical support;
* patients undergoing combined surgery;
* patients undergoing single aortocoronary bypass surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients with coronary artery disease and an indication for surgical revascularization (coronary artery bypass grafting) who meet the above-described inclusion and exclusion criteria will be enrolled by signing the informed consent the day before surgery.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2024-11-20 (Estimated); Primary Completion 2025-05-20 (Estimated); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
LIMA>LAD Pulsatility index (PI) modification | During the surgery, out of cardiopulmonary bypass
  The primary aim of this study is to assess whether a graft for a non-LAD coronary target modifies the performance (measured by flowmetry) of the flow in the LIMA>LAD graft.
  PI is expressed by the ratio of the flow volume amplitude and mean flow volume, both quantified by a flowmeter (ml/min / ml/min). An ideal value would be < 3

SECONDARY OUTCOMES:
LIMA>LAD mean flow change | During surgery, before and after transient occlusion of the other grafts for non-LAD coronary targets
  under rest conditions and after pharmacological stress. The unit of measure will be ml/min. The average flow should be above 20 ml/min.
LIMA>LAD Diastolic filling (%DF) change | During surgery,before and after transient occlusion of the other grafts for non-LAD coronary targets.
  under rest conditions and after pharmacological stress. The unit of measure will be the ratio between two parameters expressed by ml/min.
variation of Diastolic filling (%DF) on the right coronary | During surgery,before and after transient occlusion of the other grafts for non-LAD coronary targets.
  depending on its dominance or hyperdominance. The unit of measure will be the ratio between two parameters expressed by ml/min. DF% is accepted around 50%.
LIMA>LAD % Backward flow (BF) change | During surgery, before and after transient occlusion of the other grafts for non-LAD coronary targets.
  under rest conditions and after pharmacological stress. The unit of measure will be the ratio between two parameters expressed by ml/min. The identified cut-off is 3% of the total flow.
mean flow, Pulsatility Index, Diastolic filling (%DF) and Diastolic filling (%DF) in the non-LAD grafts | During surgery, before and after transient occlusion of the LIMA>LAD graft
  under rest conditions and after pharmacological stress. The meaf low will be measured in "ml/min". The others will be expressed by the ratio between two parameters expressed by ml/min.

CONTACTS AND LOCATIONS:
Overall Officials: federico cammertoni, Principal Investigator — Fondazione Policlinico Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Patient data (personal data, anthropometric data, cardiovascular risk factors, co-patologies, cardiac history, blood tests, drug therapy, electrocardiogram, echocardiogram, angiography) will be recorded

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-04): https://cdn.clinicaltrials.gov/large-docs/62/NCT06471062/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-16): https://cdn.clinicaltrials.gov/large-docs/62/NCT06471062/ICF_001.pdf